CLINICAL TRIAL: NCT07002775
Title: Use Transesophageal Echocardiography Comparing Head Up And Supine Cardiopulmonary Resuscitation On Cerebral And Systemic Hemodynamics In OHCA Patients
Brief Title: Which Position Is Better For CPR In OHCA Patients?
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202410141RINA
Record Dates: First submitted 2025-05-06; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest (CA)
Keywords: OHCA; TEE
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPR position (Other): Same patient with different CPR position : head up or supine
  Interventions: Device: Transesophageal ultrasound

INTERVENTIONS:
Device: Transesophageal ultrasound — Transesophageal ultrasound with built-in ultrasound software (Philips QLAB 3D quantification advance, Philips Healthcare, USA, speckle tracking echocardiography (STE,Speckle tracking echocardiography) to evaluate stroke volume and cardiac output in different position with the same person

SUMMARY:
Use Transesophageal ultrasound in OHCA patients to identify the proper CPR position

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest patients

Exclusion Criteria:

* DNR was signed,
* Age under 18
* Trauma patients
* Patients hard to establish advanced airway
* C spine injury patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2027-01-23 (Estimated)

PRIMARY OUTCOMES:
cardiac output | check cardiac output while CPR(Periprocedural)(after TEE insertion) in head up and supine position
  built-in ultrasound software (Philips QLAB 3D quantification advance, Philips Healthcare, USA, speckle tracking echocardiography (STE,Speckle tracking echocardiography)
stroke volume | check stroke volume while CPR(Periprocedural)(after TEE insertion) in head up and supine position
  built-in ultrasound software (Philips QLAB 3D quantification advance, Philips Healthcare,

CONTACTS AND LOCATIONS:
Overall Officials: WANCHING LIEN, Study Director — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Chang Bing Show Chawan Memorial Hospital, Changhua
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Moore JC, Salverda B, Lick M, Rojas-Salvador C, Segal N, Debaty G, Lurie KG. Controlled progressive elevation rather than an optimal angle maximizes cerebral perfusion pressure during head up CPR in a swine model of cardiac arrest. Resuscitation. 2020 May;150:23-28. doi: 10.1016/j.resuscitation.2020.02.023. Epub 2020 Feb 27. PMID 32114071
- [Background] Moore JC, Holley J, Segal N, Lick MC, Labarere J, Frascone RJ, Dodd KW, Robinson AE, Lick C, Klein L, Ashton A, McArthur A, Tsangaris A, Makaretz A, Makaretz M, Debaty G, Pepe PE, Lurie KG. Consistent head up cardiopulmonary resuscitation haemodynamics are observed across porcine and human cadaver translational models. Resuscitation. 2018 Nov;132:133-139. doi: 10.1016/j.resuscitation.2018.04.009. Epub 2018 Apr 24. PMID 29702188
- [Background] Kim T, Shin SD, Song KJ, Park YJ, Ryu HH, Debaty G, Lurie K, Hong KJ. The effect of resuscitation position on cerebral and coronary perfusion pressure during mechanical cardiopulmonary resuscitation in porcine cardiac arrest model. Resuscitation. 2017 Apr;113:101-107. doi: 10.1016/j.resuscitation.2017.02.008. Epub 2017 Feb 16. PMID 28215591
- [Background] Debaty G, Shin SD, Metzger A, Kim T, Ryu HH, Rees J, McKnite S, Matsuura T, Lick M, Yannopoulos D, Lurie K. Tilting for perfusion: head-up position during cardiopulmonary resuscitation improves brain flow in a porcine model of cardiac arrest. Resuscitation. 2015 Feb;87:38-43. doi: 10.1016/j.resuscitation.2014.11.019. Epub 2014 Nov 28. PMID 25447353